CLINICAL TRIAL: NCT06713824
Title: Neoadjuvant Radiotherapy Before Surgery for Rectal Cancer, Surgical and Oncological Outcome Analysis, Retrospective Case Control Study in a Single Institute.
Status: Active, not recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE24540A
Record Dates: First submitted 2024-11-28; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: General Surgery; Radiology
Keywords: neo-adjuvant; rectal cancer; radiotherapy; concurrent chemo-radiation therapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- neo-adjuvant radiotherapy and surgery: receive radiation therapy before surgery

SUMMARY:
Pre-operative radiotherapy for clinical stage 3 rectal cancer outcome analysis, retrospective case-control study.

DETAILED DESCRIPTION:
For clinical T3 rectal cancer, neo-adjuvant radiotherapy was proved to reduce local recurrent rate in the clinical trials. In this study, we analysis surgical and oncological outcomes of neo-adjuvant radiotherapy for stage 3 rectal cancer in the real world in a single institute and do further subgroups analysis as references for treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer, clinical stage T3 or higher, with no distant metastasis.
* Age > =20 years, ASA class I-III.
* Underwent surgery.
* Complete medical records.

Exclusion Criteria:

* Non-rectal cancer.
* Clinical stage T1-T2.
* Stage IV with distant metastasis.
* Age < 20 years, ASA class IV-V.
* Incomplete medical records.
* HIV-positive patients (Human Immunodeficiency Virus).
* Patients who completed treatment after October 1, 2024.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study collected clinical stage 3 rectal cancer patients who underwent radical resection without neoadjuvant radiotherapy at Taichung Veterans General Hospital from January 1, 2017 to October 1, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 5-year postoperative period
  The disease recurrence rate refers to the likelihood of a disease reappearing after initial treatment, encompassing both local recurrence and distant metastasis.
  Local recurrence is defined by medical standards as the reappearance of a tumor at the original site or nearby lymph nodes, typically confirmed through imaging or pathological examination and commonly occurring within 1-3 years post-surgery.
  Distant metastasis, on the other hand, is identified when tumor cells spread to distant organs, such as the liver, lungs, or bones, and is confirmed through imaging modalities (e.g., CT, MRI, or PET scans) or biopsy. The incidence of distant metastasis is closely related to tumor staging, such as the TNM classification.
survival rate | 5-year postoperative period
  This refers to the percentage of patients who are alive at a certain point in time after treatment, often 5 years, from diagnosis or start of treatment. The 5-year survival rate is commonly used in cancer research.

SECONDARY OUTCOMES:
Complication rate | 30 days after surgery
  Complications are common during post-operative treatment. Complication rate is the proportion of patients who experience an adverse event or secondary health problem as a result of the disease or the treatment provided. Some common complications include intestinal obstruction, wound infection, pneumonia, anastomotic fistula, chylous leak, and urinary tract infection (UTI).
Complications of radiation and chemotherapy | 30 days after radiation and chemotherapy
  Radiation and chemotherapy are essential cancer treatments but come with potential complications. Common radiation-related complications include skin reactions, fatigue, nausea, pulmonary toxicity, and bowel/bladder issues. Chemotherapy can lead to myelosuppression, nausea, alopecia, mucositis, and neuropathy. Measures to manage these complications include supportive care, prophylactic medications (e.g., antiemetics, growth factors), and close monitoring. Standards such as the CTCAE and Clavien-Dindo classification are used to assess and report the severity of adverse events. Personalized treatment plans, early intervention, and patient education are key to minimizing risks and improving patient outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan